CLINICAL TRIAL: NCT06707077
Title: The Effect of Sevoflurane on Cardiac Output, Mean Systemic Filling Pressure, and Vascular Resistances in Children
Brief Title: The Effect of Sevoflurane on Haemodynamics
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: HL-002-2024
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Sevoflurane; Cardiac Output; Venous Return; Vascular Resistance
Keywords: sevoflurane; cardiac output; mean systemic filling pressure; vascular resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exposure: The patient receives three increasing target end-tidal concentrations of sevoflurane, depending on what is hemodynamically (i.e. arterial hypotension) feasible in the individual patient.

SUMMARY:
Cardiac output (CO) is measured using Mostcare. Mean systemic filling pressure (MSFP) and vascular resistances are calculated using venous return curves constructed by measuring steady-state arterial and venous pressures and cardiac output (CO) during inspiratory hold manoeuvres at increasing plateau pressures. Measurements are performed at three incremental levels of targeted sevoflurane concentrations.

DETAILED DESCRIPTION:
Tracheal intubation is performed after anesthesia induction with sevoflurane. Radial arterial is cannulated and pressure transducer is connected to MostCare (core technique PRAM). HR, MAP, CVP, CO, SVR, PPV, and dp/dt are recorded at three incremental levels of targeted sevoflurane concentrations. MSFP and vascular resistances are calculated.

ELIGIBILITY:
Inclusion Criteria:

* American Association of Anesthesiologists (ASA)physical status score I-III
* major elective surgery that dictates the use of invasive hemodynamic monitoring including CVP and continuous arterial blood pressure monitoring.

Exclusion Criteria:

* symptomatic peripheral vascular disease or pulmonary disease
* aberrant cardiovascular anatomy
* significant valvular regurgitation
* severe arrhythmia

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study enrolls patients 3-10 years, with American Association of Anesthesiologists (ASA) physical status score I-III, scheduled for major elective surgery that dictates the use of invasive hemodynamic monitoring including CVP and continuous arterial blood pressure monitoring. Patients with symptomatic peripheral vascular disease or pulmonary disease, aberrant cardiovascular anatomy, significant valvular regurgitation, or severe arrhythmias are excluded.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
cardiac output | Hemodynamic parameters are recorded after 15 min of equilibration at each sevoflurane concentration.
  Cardiac output is monitored using Mostcare via a radial arterial catheter connected to the pressure transducer.
mean systemic filling pressure | Hemodynamic parameters are recorded after 15 min of equilibration at each sevoflurane concentration.
  Mean systemic filling pressure (MSFP) is calculated using venous return curve constructed by measuring steady-state arterial and venous pressures and CO during inspiratory hold manoeuvres at increasing plateau pressures. The CVP and CO data are fitted by linear regression to define the venous return curve. We define MSFP by extrapolation to zero flow.
vascular resistance | Hemodynamic parameters are recorded after 15 min of equilibration at each sevoflurane concentration.
  Total systemic vascular resistance (Rsys) is calculated as the ratio of the pressure difference between mean Pa and mean CVP and CO. The resistance downstream to MSFP is taken to reflect the resistance to venous return (Rv) and is calculated as the ratio of the pressure difference between MSFP and CVP and CO. Systemic arterial resistance (Ra) is taken to be the difference between systemic and venous resistance.

SECONDARY OUTCOMES:
mean arterial pressure | Hemodynamic parameters are recorded after 15 min of equilibration at each sevoflurane concentration.
  Systemic arterial blood pressure is monitored via a radial arterial catheter connected to a pressure transducer.
central venous pressure | Hemodynamic parameters are recorded after 15 min of equilibration at each sevoflurane concentration.
  CVP is measured with a catheter inserted through the right internal jugular vein.
pulse pressure variation | Hemodynamic parameters are recorded after 15 min of equilibration at each sevoflurane concentration.
  PPV is obtained from Mostcare.
dP/dt | Hemodynamic parameters are recorded after 15 min of equilibration at each sevoflurane concentration.
  dP/dt is obtained from Mostcare.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Wang, MD, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan university, Shanghai, China